CLINICAL TRIAL: NCT00860314
Title: Prospective, Randomized Single-center Study for Efficacy of Antero-posterior and Antero-lateral Electrode Position for External Electrical Cardioversion of Typical Atrial Flutter
Brief Title: Antero-posterior Versus Antero-lateral Electrode Position for Electrical Cardioversion of Typical Atrial Flutter
Acronym: APOVERSAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Statistical interim analysis showed valid and significant results
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stephan Willems, Ltd. Oberarzt des Universitären Herzzentrums Hamburg, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKE-2383
Record Dates: First submitted 2008-11-10; First posted 2009-03-12 (Estimated); Results first posted 2009-03-12 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Atrial Flutter
Keywords: external electrical cardioversion; typical atrial flutter; electrode position; antero-lateral; antero-posterior; biphasic cardioversion; step-up protocol
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AP Position (Active Comparator): Cardioversion with antero-posterior electrode position
  Interventions: Procedure: external electrical cardioversion (with antero-posterior electrode position)
- AL Position (Active Comparator): Cardioversion with antero-lateral electrode position
  Interventions: Procedure: external electrical cardioversion (with antero-lateral electrode position)

INTERVENTIONS:
Procedure: external electrical cardioversion (with antero-posterior electrode position) — external biphasic electrical cardioversion with step-up-protocol of 50-75-100-150-200 Joules if necessary with antero-posterior electrode position until restoration of normal sinus rhythm
  Other Names: biphasic cardioversion; countershock treatment
  Arms: AP Position
Procedure: external electrical cardioversion (with antero-lateral electrode position) — external biphasic electrical cardioversion with step-up protocol of 50-75-100-150-200 Joules if necessary with antero-lateral electrode position until restoration of normal sinus rhythm
  Other Names: biphasic cardioversion; countershock treatment
  Arms: AL Position

SUMMARY:
The aim of this study is to identify the one electrode position out of two most commonly used for external electrical cardioversion of typical atrial flutter, which needs less delivered energy and less needed number of shocks for successful cardioversion.

DETAILED DESCRIPTION:
Typical atrial flutter is the second-most prevalent atrial tachyarrhythmia. No guidelines for treatment exist and few studies investigate treatment of atrial flutter. Mostly, guidelines for atrial fibrillation are followed for treatment of atrial flutter. Atrial flutter has a different pathomechanism as atrial fibrillation, therefore special guidelines for treatment are needed. Among drug treatment and ablation procedures, external electrical cardioversion is commonly used, especially for treatment of acute symptomatic patients. This study may help to further define safe and successful procedures for electrical cardioversion of atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of typical atrial flutter
* signed written informed consent
* eligibility for sedation and external electrical cardioversion

Exclusion Criteria:

* clinical diagnosis of arrhythmia other than typical atrial flutter
* implanted ICD or pacemaker
* proof of atrial thrombi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, Prof. Dr., Study Chair — Oberarzt
Locations (1):
- University Hospital Hamburg-Eppendorf, Heart Center, Hamburg, Germany

REFERENCES:
- [Background] Kerber RE, Kouba C, Martins J, Kelly K, Low R, Hoyt R, Ferguson D, Bailey L, Bennett P, Charbonnier F. Advance prediction of transthoracic impedance in human defibrillation and cardioversion: importance of impedance in determining the success of low-energy shocks. Circulation. 1984 Aug;70(2):303-8. doi: 10.1161/01.cir.70.2.303. PMID 6733884
- [Background] Kirchhof P, Eckardt L, Loh P, Weber K, Fischer RJ, Seidl KH, Bocker D, Breithardt G, Haverkamp W, Borggrefe M. Anterior-posterior versus anterior-lateral electrode positions for external cardioversion of atrial fibrillation: a randomised trial. Lancet. 2002 Oct 26;360(9342):1275-9. doi: 10.1016/s0140-6736(02)11315-8. PMID 12414201
- [Background] Kirchhof P, Borggrefe M, Breithardt G. Effect of electrode position on the outcome of cardioversion. Card Electrophysiol Rev. 2003 Sep;7(3):292-6. doi: 10.1023/B:CEPR.0000012399.96959.ab. PMID 14739731
- [Background] Kerber RE, Jensen SR, Grayzel J, Kennedy J, Hoyt R. Elective cardioversion: influence of paddle-electrode location and size on success rates and energy requirements. N Engl J Med. 1981 Sep 17;305(12):658-62. doi: 10.1056/NEJM198109173051202. PMID 7266602
- [Background] Botto GL, Politi A, Bonini W, Broffoni T, Bonatti R. External cardioversion of atrial fibrillation: role of paddle position on technical efficacy and energy requirements. Heart. 1999 Dec;82(6):726-30. doi: 10.1136/hrt.82.6.726. PMID 10573502
- [Background] Yoon RS, DeMonte TP, Hasanov KF, Jorgenson DB, Joy ML. Measurement of thoracic current flow in pigs for the study of defibrillation and cardioversion. IEEE Trans Biomed Eng. 2003 Oct;50(10):1167-73. doi: 10.1109/TBME.2003.816082. PMID 14560770
- [Background] Van Gelder IC, Tuinenburg AE, Schoonderwoerd BS, Tieleman RG, Crijns HJ. Pharmacologic versus direct-current electrical cardioversion of atrial flutter and fibrillation. Am J Cardiol. 1999 Nov 4;84(9A):147R-151R. doi: 10.1016/s0002-9149(99)00715-8. PMID 10568674
- [Background] Kerber RE. Transthoracic cardioversion of atrial fibrillation and flutter: standard techniques and new advances. Am J Cardiol. 1996 Oct 17;78(8A):22-6. doi: 10.1016/s0002-9149(96)00562-0. PMID 8903272
- [Background] Camacho MA, Lehr JL, Eisenberg SR. A three-dimensional finite element model of human transthoracic defibrillation: paddle placement and size. IEEE Trans Biomed Eng. 1995 Jun;42(6):572-8. doi: 10.1109/10.387196. PMID 7790013
- [Background] Kirchhof P, Monnig G, Wasmer K, Heinecke A, Breithardt G, Eckardt L, Bocker D. A trial of self-adhesive patch electrodes and hand-held paddle electrodes for external cardioversion of atrial fibrillation (MOBIPAPA). Eur Heart J. 2005 Jul;26(13):1292-7. doi: 10.1093/eurheartj/ehi160. Epub 2005 Feb 25. PMID 15734772
- See also: Homepage of University Hospital Hamburg-Eppendorf — http://www.uke.de

RESULTS

PARTICIPANT FLOW:
Groups:
- Antero-Posterior Group: Cardioversion with antero-posterior electrode position
- Antero-Lateral Group: Cardioversion with antero-lateral electrode position
Period: Overall Study
Arm/Group | Antero-Posterior Group | Antero-Lateral Group
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antero-Posterior Group | Antero-Lateral Group | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 31 | 58
  >=65 years | 21 | 17 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12.18) | 62 (12.53) | 62 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 37 | 35 | 72
Region of Enrollment [Number; unit: participants]
  Germany | 48 | 48 | 96

OUTCOME MEASURES:

1. Secondary Outcome: Mean Number of Cardioversion Shocks
Time Frame: 30 seconds after cardioversion
Measure: Mean (Standard Deviation); unit: Shocks
Arm/Group | Antero-Posterior Group | Antero-Lateral Group
Number analyzed (Participants) | 48 | 48
Shocks | 1.96 (1.00) | 1.48 (1.01)

2. Primary Outcome: Number of Successfully Cardioverted Participants for Each Electrode Position
Description: After restoration of normal sinus rhythm for 30 seconds and longer by electrical countershock a cardioversion is counted as successful.
Time Frame: 30 seconds after cardioversion
Measure: Number; unit: participants
Arm/Group | Antero-Posterior Group | Antero-Lateral Group
Number analyzed (Participants) | 48 | 48
participants | 48 | 48

3. Secondary Outcome: Mean Energy Requirement for Successful Cardioversion
Description: Overall energy in the mean (number of joules) necessary for successful cardioversion of all patients per group.
Time Frame: 30 seconds after cardioversion
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | Antero-Posterior Group | Antero-Lateral Group
Number analyzed (Participants) | 48 | 48
Joules | 77 (13) | 65 (13)

4. Secondary Outcome: Number of Participants Succesfully Cardioverted With First Shock in Each Electrode Position
Description: Number of participants successfully cardioverted to normal sinus rhythm with one shock of 50 Joules.
Time Frame: 30 seconds after cardioversion
Measure: Number; unit: participants
Arm/Group | Antero-Posterior Group | Antero-Lateral Group
Number analyzed (Participants) | 48 | 48
participants | 17 | 35

ADVERSE EVENTS:
Arm/Group | Antero-Posterior Group | Antero-Lateral Group
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes